CLINICAL TRIAL: NCT01387204
Title: An Open-label Mass Balance Study to Investigate the Absorption, Distribution, Metabolism and Elimination of a Single Oral Dose of MEK Inhibitor [14C]GSK1120212 in Male Subjects With Solid Tumors
Brief Title: Study to Investigate the Absorption, Distribution, Metabolism and Elimination of [14C]GSK1120212
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113708
Record Dates: First submitted 2011-06-09; First posted 2011-07-04 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: MEK inhibitor; elimination; Phase 1; GSK1120212; cancer; Pharmacokinetics; oncology; radiolabeled ADME
MeSH Terms: conditions — Neoplasms | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-Dose, 2 mg [14C]GSK1120212 (Experimental): A single 2 mg (2 mg/10mL) oral dose of [14C]GSK1120212 containing approximately 79 μCi of radioactivity will be delivered as a solution.
  Interventions: Drug: GSK1120212

INTERVENTIONS:
Drug: GSK1120212 — The 2 mg dose is based on clinical data from the ongoing FTIH study in which subjects have been dosed daily for greater than 21 days, as well as preclinical toxicity data.

SUMMARY:
GSK1120212 is a reversible and highly selective allosteric inhibitor of MEK1 and MEK2 activation and kinase activity currently being developed for the treatment of malignant melanoma. This is a Phase I, open-label, non-randomized, single-dose study designed to characterize the absorption, distribution, metabolism, and elimination (ADME) of a single oral dose of MEK inhibitor [14C]GSK1120212 as a solution in male subjects with solid tumor malignancies. A sufficient number of subjects will be enrolled to complete approximately four evaluable subjects. Following completion of the study, subjects may elect to continue dosing with GSK1120212 in the rollover study, MEK114375.

ELIGIBILITY:
Inclusion Criteria:

1. Male 18 years old or older.
2. Written informed consent provided
3. Body weight greater than or equal to 45 kg and a BMI greater than or equal to 19 kg/m2 and less than or equal to 35 kg/m2 (inclusive).
4. Able to swallow and retain oral medication.
5. Histologically or cytologically confirmed diagnosis of a solid tumor.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
7. Agree to use one of the contraception methods listed in the protocol from the time of the first dose of study medication until sixteen weeks after the last dose of study medication.
8. A history of regular bowel movements (approximately once per day).
9. Adequate baseline organ function as listed in the protocol.

Exclusion Criteria:

1. Currently receiving cancer therapy as specified in the protocol.
2. Serious and/or unstable pre-existing medical psychiatric disorder, or other conditions.
3. Any major surgery within the last four weeks.
4. Unresolved toxicity equal to or greater than Grade 2 from previous anti-cancer therapy except alopecia.
5. An occupation within the past 12 months which requires monitoring for radiation exposure, nuclear medicine procedures or excessive x-rays.
6. Radiation exposure from the previous three year period over 10 mSv if exposed to ionizing radiation above background as a result of work with radiation as category A (classified) workers or as a result of research studies.
7. History of interstitial lung disease or pneumonitis.
8. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to dimethyl sulfoxide (DMSO).
9. Current use of a prohibited medications described in the protocol.

   • Use of anticoagulants such as warfarin is permitted.
10. History RVO or CSR.

    * Predisposing factors to RVO or CSR.
    * Visible retinal pathology that is considered a risk factor for RVO or CSR such as:

      - Evidence of new optic disc cupping

      - Intraocular pressure greater than 21 mm Hg as measured by tonography. 11.1. Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression. (Previously treated and have had stable CNS disease for greater than 3 months, asymptomatic and off corticosteroids, or on stable dose of corticosteroids for at least 1 month prior to study Day 1 are permitted).

11.2. Receiving enzyme inducing anti-epileptic drugs (EIAEDs). 12. History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within the past 6 months. 13. QTcB greater than or equal to 480 msec. 14. History or evidence of current clinically significant uncontrolled arrhythmias.

15. History or evidence of current greater than or equal to Class II congestive heart failure.

16. Active gastrointestinal disease or other condition (e.g., gastrectomy, bariatric surgery, small bowel or large bowel resection, or cholecystectomy).

17. A history of known Human Immunodeficiency Virus (HIV), Hepatitis B Virus, or Hepatitis C Virus.

18. Alcohol or drug abuse within six months prior to screening. 19. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drugs or excipients.

20. Participated in a clinical trial and has received an investigational product within 30 days or five half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) before the 1st dose.

21. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.

22. Mentally or legally incapacitated.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-02-15 (Actual); Primary Completion 2011-07-18 (Actual); Study Completion 2011-07-18 (Actual)

PRIMARY OUTCOMES:
Total excretion of radioactivity | 11 days
  • Total and relative excretion of radioactivity in urine and feces following a single, 2 mg oral solution dose of [14C]GSK1120212

SECONDARY OUTCOMES:
Total radioactivity concentration in blood and plasma | 11 days
  AUC(0- t), AUC(0-∞), Cmax, tmax and t1/2
Characterize and quantify metabolites in urine plasma and feces | 11 days
  Characterize and quantify metabolites of GSK1120212 in plasma, urine and feces (studied separately under a DMPK protocol).
Assess covalent binding of drug related material to plasma proteins | 11 days
  Assess percentage of drug-related material that covalently bonds to plasma proteins (studied separately under a DMPK protocol)
Blood:plasma ratio | 11 days
  Blood:plasma ratio of total drug-related material (radioactivity)
Pharmacokentic concentrations in plasma | 11 days
  Plasma GSK1120212 concentrations AUC(0-t), AUC(0-∞), Cmax, tmax, and t1/2
AEs | From dosing on Day 1 to Follow-up
  Number of adverse events (AEs)
Vital signs | Screening, Day -1, Day 1, Day 5, and Follow-up
  Changes from baseline
ECGs | Screening, Day 1 pre-dose, 24 hours, Day 11 and Follow-up
  Changes from baseline
Clinical Laboratory assessments | Screening, Day -1, and Day 11
  Changes from baslines

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tacoma, Washington, United States

REFERENCES:
- [Background] Allen LF, Sebolt-Leopold J, Meyer MB. CI-1040 (PD184352), a targeted signal transduction inhibitor of MEK (MAPKK). Semin Oncol. 2003 Oct;30(5 Suppl 16):105-16. doi: 10.1053/j.seminoncol.2003.08.012. PMID 14613031
- [Background] Davies H, Bignell GR, Cox C, Stephens P, Edkins S, Clegg S, Teague J, Woffendin H, Garnett MJ, Bottomley W, Davis N, Dicks E, Ewing R, Floyd Y, Gray K, Hall S, Hawes R, Hughes J, Kosmidou V, Menzies A, Mould C, Parker A, Stevens C, Watt S, Hooper S, Wilson R, Jayatilake H, Gusterson BA, Cooper C, Shipley J, Hargrave D, Pritchard-Jones K, Maitland N, Chenevix-Trench G, Riggins GJ, Bigner DD, Palmieri G, Cossu A, Flanagan A, Nicholson A, Ho JW, Leung SY, Yuen ST, Weber BL, Seigler HF, Darrow TL, Paterson H, Marais R, Marshall CJ, Wooster R, Stratton MR, Futreal PA. Mutations of the BRAF gene in human cancer. Nature. 2002 Jun 27;417(6892):949-54. doi: 10.1038/nature00766. Epub 2002 Jun 9. PMID 12068308
- [Background] GlaxoSmithKline Document Number HM2009/00151/01 GSK1120212 Investigator's Brochure Report Date 4 June 2010.
- [Background] GlaxoSmithKline Document Number RD2009/01379/00. Dosimetry Review for oral [14C]GSK1120212. Report Date 19-Nov-2009.
- [Background] GlaxoSmithKline Document Number RM2007/00642/03. MEK111054: An open-label, multiple-dose, dose escalation study to investigate the safety, harmacokinetics, and pharmacodynamics of the MEK inhibitor GSK1120212 in subjects with solid tumors or lymphoma. 2009.
- [Background] Lorusso PM, Adjei AA, Varterasian M, Gadgeel S, Reid J, Mitchell DY, Hanson L, DeLuca P, Bruzek L, Piens J, Asbury P, Van Becelaere K, Herrera R, Sebolt-Leopold J, Meyer MB. Phase I and pharmacodynamic study of the oral MEK inhibitor CI-1040 in patients with advanced malignancies. J Clin Oncol. 2005 Aug 10;23(23):5281-93. doi: 10.1200/JCO.2005.14.415. Epub 2005 Jul 11. PMID 16009947
- [Background] LoRusso PM, Krishnamurthi S, Rinehart JR, et al. A Phase 1-2 clinical study of the second-generation MEK inhibitor, PD 0325901 in patients with advanced cancer. J Clin Oncol. 2005; 23:3011.
- [Background] LoRusso PM, Krishnamurthi SS, Rinehart JJ, Nabell LM, Croghan GA, Chapman PB, Selaru P, Kim S, Ricart AD, Wilner KD. Clinical aspects of a phase I study of PD-0325901, a selective oral MEK inhibitor, in patients with advanced cancer. Presented at AACR-NCI-EORTC International Conference on Molecular Targets and Cancer Therapeutics 2007; 6:3649s [abstr B113].
- [Background] NCI. Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. DHHS,NCI, NIH, Bethesda, MD; 2009.
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Tzekova, V, Cebotaru C, Ciuleanu TE, et al. Efficacy and safety of AZD6244 (ARRY-142886) as second/third-line treatment of patients (pts) with advanced non-small cell lung cancer (NSCLC). J Clin Oncol. 2008; 26:431s.
- See also: Results for study 113708 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113708?search=study&search_terms=113708#rs